CLINICAL TRIAL: NCT00832221
Title: An Open Label, 1-sequence Cross-over, Positron Emission Tomography (PET) Study With [11C]Raclopride to Determine Central D2 Dopamine Receptor Occupancy of Quetiapine Fumarate Immediate Release (SEROQUEL®) With Quetiapine Fumarate Extended Release (SEROQUEL XR®) in Healthy Male Volunteers
Brief Title: Positron Emission Tomography (PET) Study With [11C]Raclopride to Determine Central D2 Dopamine Occupancy of SEROQUEL
Acronym: PET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Märta Segerdahl, MD, PhD, Medical Science Director, Clinical Discovery Team, AstraZeneca
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D1443C00038; EudractCT 2008-006553-40
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2009-09-14 (Estimated); Status verified 2009-09

CONDITIONS: Depression
Keywords: PET; Phase 1; Depression; SEROQUEL; Positron Emission Tomography; Drug profile comparison
MeSH Terms: conditions — Depression | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: SEROQUEL XR (quetiapine); Drug: radioligand [11C]raclopride
- 2 (Active Comparator)
  Interventions: Drug: SEROQUEL IR (quetiapine); Drug: radioligand [11C]raclopride

INTERVENTIONS:
Drug: SEROQUEL XR (quetiapine) — repeated dose of oral tablets, 8 times per subject
  Arms: 1
Drug: SEROQUEL IR (quetiapine) — repeated dose of oral tablets, 4 times per subject
  Arms: 2
Drug: radioligand [11C]raclopride — single dose of iv admin, 5 times per subject

SUMMARY:
The aim of this study is to relate pharmacokinetics of two different formulations of quetiapine to PET measured receptor occupancy in the brains of healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Normal MRI scan
* Body mass index 19-30 kg/m2 and weight of 50-100 kg
* Clinically normal physical findings, medical history and laboratory values

Exclusion Criteria:

* Trauma or sickness last 2 weeks before the first PET examination.
* A history or presence of neurological, haematological, psychiatric, gastrointestinal, hepatic, pulmonary, renal disease or other condition as judged by the Investigator
* Any previous participation in a PET study
* Subjects suffer from claustrophobia

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-01; Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Positron emission tomography using the radioligand [11C]raclopride | 5 visits

SECONDARY OUTCOMES:
Adverse Events (AEs), vital signs and changes in laboratory parameters, physical examinations, Alertness Visual Analogue Scale. | 5 visits. Some tests will be done several times per visit. All tests will not be performed at every visit.
Pharmacokinetics of quetiapine and its main active metabolite | 22 samples

CONTACTS AND LOCATIONS:
Overall Officials: Ingemar Bylesjö, MD, PhD, Principal Investigator — AstraZeneca Clinical Pharmacology Unit, Stockholm, Sweden; Sophia Bengtsson, Study Director — AstraZeneca R&D, Södertälje, Sweden
Locations (1):
- Research Site, Stockholm, Sweden

REFERENCES:
- [Derived] Nord M, Nyberg S, Brogren J, Jucaite A, Halldin C, Farde L. Comparison of D(2) dopamine receptor occupancy after oral administration of quetiapine fumarate immediate-release and extended-release formulations in healthy subjects. Int J Neuropsychopharmacol. 2011 Nov;14(10):1357-66. doi: 10.1017/S1461145711000514. Epub 2011 Apr 11. PMID 21477416